CLINICAL TRIAL: NCT04907084
Title: Phase 2a Study of the Effect of Serine Supplementation and Fenofibrate Treatment on Serum Deoxysphinganine Levels in Patients With Macular Telangiectasia (MacTel) Type 2 (SAFE Study)
Brief Title: Serine and Fenofibrate Study in Patients With MacTel Type 2
Acronym: SAFE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2020-002
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Macular Telangiectasia Type 2
MeSH Terms: interventions — Serine; Fenofibrate

STUDY DESIGN:
Intervention Model Description: The randomization model will stratify patients by diabetes status, ensuring equal treatment of diabetics / non-diabetics in the study. A permuted block design will be used to randomize participants in a 1:1:1:1:1:1 ratio to either 1) serine 200 mg/kg/day, 2) serine 400 mg/kg/day, 3) fenofibrate 200 mg/day, 4) serine 200 mg/kg/day AND fenofibrate 200 mg/day, 5) serine 400 mg/kg/day AND fenofibrate 200 mg/day, or 6) no treatment (control group).
Masking Description: This is an open-label study. Participants will be told if they are taking serine and/or fenofibrate, or if they are participating as a control (no treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Serine 200 mg/kg/day (Experimental): Serine 200 mg/kg per day. To be taken once per day for 6 weeks. Exact dose dependent on participant's weight (in kg)).
  Interventions: Dietary Supplement: Serine
- Serine 400 mg/kg/day (Experimental): Serine 400 mg/kg per day. To be taken once per day for 6 weeks. Exact dose dependent on participant's weight (in kg)).
  Interventions: Dietary Supplement: Serine
- Fenofibrate 160 mg/day (Experimental): Fenofibrate 160 mg per day. To be taken once per day for 6 weeks.
  Interventions: Drug: Fenofibrate
- Serine 200 mg/kg/day and Fenofibrate 160 mg/day (Experimental): Serine 200 mg/kg per day. To be taken once per day for 6 weeks. Exact dose dependent on participant's weight (in kg)).
  Fenofibrate 160 mg per day. To be taken once per day for 6 weeks.
  Interventions: Dietary Supplement: Serine; Drug: Fenofibrate
- Serine 400 mg/kg/day and Fenofibrate 160 mg/day (Experimental): Serine 400 mg/kg per day. To be taken once per day for 6 weeks. Exact dose dependent on participant's weight (in kg)).
  Fenofibrate 160 mg per day. To be taken once per day for 6 weeks.
  Interventions: Dietary Supplement: Serine; Drug: Fenofibrate
- No treatment (No Intervention): Control group: no investigational product taken

INTERVENTIONS:
Dietary Supplement: Serine — Powdered serine supplement (Dosed out individually per participant. Participant to mix with water and ingest orally)
  Arms: Serine 200 mg/kg/day; Serine 200 mg/kg/day and Fenofibrate 160 mg/day; Serine 400 mg/kg/day; Serine 400 mg/kg/day and Fenofibrate 160 mg/day
Drug: Fenofibrate — Fenofibrate 160mg pill, taken orally
  Arms: Fenofibrate 160 mg/day; Serine 200 mg/kg/day and Fenofibrate 160 mg/day; Serine 400 mg/kg/day and Fenofibrate 160 mg/day

SUMMARY:
This is a Phase 2a study of the effect of serine supplementation and fenofibrate treatment on serum deoxysphingolipid levels in patients with macular telangiectasia type 2 (MacTel). This study involves six arms. Participants will be randomly assigned to one of the following treatment groups: serine 200 mg/kg/day, serine 400 mg/kg/day, fenofibrate 160 mg/day, both serine 200 mg/kg/day and fenofibrate 160 mg/day, both serine 400 mg/kg/day and fenofibrate 160 mg/day, or no treatment (control group). Serum deoxysphingolipid levels will be used as the primary outcome, and safety will be evaluated. The participants will be followed for 10 weeks, with visits at Screening, Week 0, 3, 6 and 10.

DETAILED DESCRIPTION:
Additional Procedures include:

1. Fasting blood work
2. Collection of microbiome samples

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent obtained from the participant in accordance with the local regulations;
2. Males/females 21 years of age or older;
3. English speaking;
4. Enrolled in the Natural History Observation and Registry Study (NHOR) and diagnosed with confirmed MacTel type 2 in at least one eye;
5. Willing to use contraception, if applicable; and
6. Willing to comply with study protocol and follow-up visits.

Exclusion Criteria:

1. Participant is unable to provide informed consent;
2. Participant is less than 21 years of age;
3. Participant is currently taking, or has taken within four weeks prior to screening, a serine or glycine supplement;
4. Participant is currently taking, or has taken within 12 months prior to screening, fibrates including clofibrate, ciprofibrate, bezafibrate, fenofibrate, and gemfibrozil;
5. Participant is currently taking an anticoagulant, colchicine, cyclosporine, tacrolimus or bile acid binding resins;
6. Participant has known allergy to fibrates and/or serine;
7. Participant has a known history of clinically significant myopathy or myalgia related to cholesterol-lowering drugs;
8. Participant has active liver disease and/or elevated liver enzymes*;
9. Participant has renal dysfunction as evidenced by elevated serum creatinine* and/ or glomerular filtration rate (GFR) less than 90 mL/min;
10. Participant has thrombocytopenia as evidenced by a platelet count below 100,000 per microliter, anemia as evidenced by hemoglobin levels below 10 g/dL, or history of bleeding disorder;
11. Participant has a history of gallbladder disease or has had a cholecystectomy;
12. Participant has triglyceride levels greater than 400 mg/dL on treatment, or greater than 700 mg/dL on no treatment;
13. Participant has untreated/uncured Hepatitis C, or a history of Hepatitis B, autoimmune hepatitis, or HIV;
14. Participant has had any malignancies within the last 5 years (not including basal cell carcinoma);
15. Participant has ever been enrolled in a clinical trial involving ciliary neurotrophic factor (CNTF) treatment;
16. Participant is currently enrolled in another clinical trial that involves treatment or participated in one within the last 30 days;
17. Participant is pregnant, breastfeeding or planning a pregnancy;
18. Participant is medically unable to comply with study procedures or follow-up visits;
19. Participant has, in the opinion of the Investigator, any physical or mental condition that would increase the patient's risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments; or
20. Patient is unavailable for follow-up visits. *based on reference range for the local laboratory used

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Serum Deosxysphingolipid Levels | blood draws from week 3, 6, and 10
  Any changes in serum deoxysphingolipid levels measured (determined via serum sample) at 3 weeks, 6 weeks, and/or 10 weeks when compared with baseline levels measured in week 0
Safety Assessment | Assessment at each study visit (reviewed at week 3, week 6, and week 10 of study)
  Safety assessment measured via examined AEs and SAEs (during study visits) and via participant self-reported AEs and SAEs that occurred between visits

SECONDARY OUTCOMES:
Lipid Levels | blood draws from week 3, 6, and 10
  Any changes in lipid levels measured (determined via blood tests) at 3 weeks, 6 weeks, and/or 10 weeks when compared with baseline levels measured at screening
Amino Acid Levels | blood draws from week 3, 6, and 10
  Any changes in amino acid levels measured (determined via blood tests) at 3 weeks, 6 weeks, and/or 10 weeks when compared with baseline levels measured at screening

CONTACTS AND LOCATIONS:
Overall Officials: Mari A Gantner, PhD, Principal Investigator — Lowy Medical Research Institute
Locations (9):
- United States (8):
  - Emory University, Atlanta, Georgia
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Moran Eye Center, University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - The Eye Institute, Medical College of Wisconsin, Milwaukee, Wisconsin
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No